CLINICAL TRIAL: NCT05558878
Title: Effect of Ambroxol on the Inflammatory Markers and Clinical Outcome of Patients With Diabetic Peripheral Neuropathy
Brief Title: Effect of Ambroxol in Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Beshoy Thabit, Clinical Pharmacy demonstrator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ambroxol in DPN
Record Dates: First submitted 2022-09-21; First posted 2022-09-28 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Neuropathy Peripheral
Keywords: Diabetic Complications; Diabetic Peripheral Neuropathy; Inflammatory markers; Tumor necrosis alpha; nuclear factor kappa-light-chain-enhancer of activated B cells; Oxidative stress; Superoxide dismutase
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambroxol (intervention arm) (Experimental): 40 patients will receive conventional therapy for diabetic neuropathy in addition to ambroxol 450 mg/day divided into 3 doses (each dose consists of 2 75mg capsules) daily for 3 months.
  Interventions: Drug: Ambroxol Oral Product
- Control arm (No Intervention): 40 patients will receive conventional therapy for diabetic neuropathy for 3 months.

INTERVENTIONS:
Drug: Ambroxol Oral Product — Drug: Ambroxol (75 mg capsule)
  Ambroxol is a mucolytic and expectorant drug. Ambroxol has been approved as lozenges for topical analgesia of sore throat in pharyngitis owing to its local anesthetic properties. Anti-inflammatory properties of ambroxol were confirmed by numerous studies. Ambroxol affect neuronal transduction by blocking (TTX)-resistant Na+ channels (Nav1.8) in small (pain-sensing) dorsal root ganglion neurons more potently than TTX-sensitive channels.
  Arms: Ambroxol (intervention arm)

SUMMARY:
A prospective, randomized, controlled study will be conducted at Department of Endocrinology, Faculty of Medicine, Ain Shams University, assessing the efficacy of Ambroxol addition on the clinical outcome and inflammatory markers in Diabetic peripheral neuropathy patients

DETAILED DESCRIPTION:
All patients presenting to the Endocrinology department, Ain Shams University Hospitals, will be assessed for eligibility as follow:

Inclusion criteria:

* Patients aged 18-75 years diagnosed with Type 2 Diabetes.
* Patients diagnosed with Peripheral Diabetic Neuropathy.

Exclusion criteria:

* Patients with autoimmune disorders (Sjogren's syndrome, lupus, rheumatoid arthritis),inherited disorders causing PN (Charcot-Marie-Tooth), thyroid diseases, patients undergone gastroplasty surgery and cancer patients.
* Pressure on or injury to the nerves
* Patients with severe kidney or liver dysfunction.
* Patients with recent history of / or ongoing infection.
* Patients with cerebral vascular disease, vasculitis, peripheral arterial disease or claudication symptoms, toxic neuritis, vitamin B12 or folate deficiency, spondyloarthropathy, foot edema or ulcer and diagnosis of other neuromuscular disorders or neurodegenerative diseases.
* Use of medications or supplements known to cause peripheral neuropathy.
* Patients consuming alcohol, any antioxidant supplements or anti-inflammatory medicines and drug abuse.
* Ketoacidosis or hypoglycemia resulting in hospital admission within the last 3 months.
* Pregnancy or lactation or expecting to get pregnant during the study.
* Medical, psychological, behavioral or pharmacological factors interfering with ability to participate in trial, collection or interpretation of study data.
* Allergy to ambroxol.

Eligible patients will be randomly assigned to one of 2 groups:

Group 1, Ambroxol group (n=40): Patients will receive conventional therapy for diabetic neuropathy in addition to ambroxol 450 mg/day divided into 3 doses (each dose consists of two 75mg tablets) daily for 3 months.

Group 2, Control group (n= 40): Patients will receive conventional therapy for diabetic neuropathy for 3 months.

All subjects will sign an informed consent statement prior to inclusion in the study.

Follow up evaluation :

All patients in both groups will be followed up every other week & will be assessed for the following:

Diabetic neuropathy scoring, occurrence of side effects & Pain assessment.

End of study evaluation :

After 3 months, all patients will be assessed for the same parameters assessed at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years diagnosed with Type 2 Diabetes.
* Patients diagnosed with Peripheral Diabetic Neuropathy.

Exclusion Criteria:

* Patients with autoimmune disorders (Sjogren's syndrome, lupus, rheumatoid arthritis),inherited disorders causing PN (Charcot-Marie-Tooth), thyroid diseases, patients undergone gastroplasty surgery and cancer patients.
* Pressure on or injury to the nerves
* Patients with severe kidney or liver dysfunction.
* Patients with recent history of / or ongoing infection.
* Patients with cerebral vascular disease, vasculitis, peripheral arterial disease or claudication symptoms, toxic neuritis, vitamin B12 or folate deficiency, spondyloarthropathy, foot edema or ulcer and diagnosis of other neuromuscular disorders or neurodegenerative diseases.
* Use of medications or supplements known to cause peripheral neuropathy.
* Patients consuming alcohol, any antioxidant supplements or anti-inflammatory medicines and drug abuse.
* Ketoacidosis or hypoglycemia resulting in hospital admission within the last 3 months.
* Pregnancy or lactation or expecting to get pregnant during the study.
* Medical, psychological, behavioral or pharmacological factors interfering with ability to participate in trial, collection or interpretation of study data.
* Allergy to ambroxol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Effect of Ambroxol on Tumor necrosis factor alpha (TNF-α) | 3 months
  Blood samples will be drawn at baseline and end of study to track changes in TNF-α using ELISA technique
Effect of Ambroxol on NF-κB (or NF-kappaB, "nuclear factor kappa-light-chain-enhancer of activated B cells") | 3 months
  Blood samples will be drawn at baseline and end of study to track changes in NF-kappaB levels using ELISA technique
Effect of Ambroxol on Superoxide dismutase | 3 months
  Blood samples will be drawn at baseline and end of study to track changes in Superoxide dismutase levels using spectrophotometric technique

SECONDARY OUTCOMES:
Effect of Ambroxol on clinical outcome : Toronto clinical scoring systems (TCSS) | 3 months
  Patient are going to be followed up every other week for detection of progression and severity of neuropathy.
Effect of Ambroxol on clinical outcome : Michigan diabetic neuropathy score (MDNS) | 3 months
  Patient are going to be followed up every other week for detection of progression and severity of neuropathy.
Effect of Ambroxol on clinical outcome : Pain assessment using the Numeric rating scale NRS | 3 months
  Patients are going to be followed up every other week to detect point decrease on pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Association, American Diabetes.
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657
- [Background] Candrilli SD, Davis KL, Kan HJ, Lucero MA, Rousculp MD. Prevalence and the associated burden of illness of symptoms of diabetic peripheral neuropathy and diabetic retinopathy. J Diabetes Complications. 2007 Sep-Oct;21(5):306-14. doi: 10.1016/j.jdiacomp.2006.08.002. PMID 17825755
- [Background] Gregg EW, Sorlie P, Paulose-Ram R, Gu Q, Eberhardt MS, Wolz M, Burt V, Curtin L, Engelgau M, Geiss L; 1999-2000 national health and nutrition examination survey. Prevalence of lower-extremity disease in the US adult population >=40 years of age with and without diabetes: 1999-2000 national health and nutrition examination survey. Diabetes Care. 2004 Jul;27(7):1591-7. doi: 10.2337/diacare.27.7.1591. PMID 15220233
- [Background] Albers JW, Pop-Busui R. Diabetic neuropathy: mechanisms, emerging treatments, and subtypes. Curr Neurol Neurosci Rep. 2014 Aug;14(8):473. doi: 10.1007/s11910-014-0473-5. PMID 24954624
- [Background] Boulton AJ, Malik RA. Diabetic neuropathy. Med Clin North Am. 1998 Jul;82(4):909-29. doi: 10.1016/s0025-7125(05)70029-8. PMID 9706126
- [Background] Soliman E,Gellido C.Diabetic Neuropathy. eMedicine.com March 29, 2002.
- [Background] Ang L, Cowdin N, Mizokami-Stout K, Pop-Busui R. Update on the Management of Diabetic Neuropathy. Diabetes Spectr. 2018 Aug;31(3):224-233. doi: 10.2337/ds18-0036. PMID 30140138
- [Background] Boulton AJ, Malik RA, Arezzo JC, Sosenko JM. Diabetic somatic neuropathies. Diabetes Care. 2004 Jun;27(6):1458-86. doi: 10.2337/diacare.27.6.1458. No abstract available. PMID 15161806
- [Background] Boulton AJ, Vinik AI, Arezzo JC, Bril V, Feldman EL, Freeman R, Malik RA, Maser RE, Sosenko JM, Ziegler D; American Diabetes Association. Diabetic neuropathies: a statement by the American Diabetes Association. Diabetes Care. 2005 Apr;28(4):956-62. doi: 10.2337/diacare.28.4.956. No abstract available. PMID 15793206
- [Background] Dyck PJ, Albers JW, Andersen H, Arezzo JC, Biessels GJ, Bril V, Feldman EL, Litchy WJ, O'Brien PC, Russell JW; Toronto Expert Panel on Diabetic Neuropathy. Diabetic polyneuropathies: update on research definition, diagnostic criteria and estimation of severity. Diabetes Metab Res Rev. 2011 Oct;27(7):620-8. doi: 10.1002/dmrr.1226. PMID 21695763
- [Background] Thomas PK. Classification, differential diagnosis, and staging of diabetic peripheral neuropathy. Diabetes. 1997 Sep;46 Suppl 2:S54-7. doi: 10.2337/diab.46.2.s54. PMID 9285500
- [Background] American Diabetes Association. Standardized measures in diabetic neuropathy. Diabetes Care 1996;19(1S):72S-92S.
- [Background] Pang L, Lian X, Liu H, Zhang Y, Li Q, Cai Y, Ma H, Yu X. Understanding Diabetic Neuropathy: Focus on Oxidative Stress. Oxid Med Cell Longev. 2020 Jul 31;2020:9524635. doi: 10.1155/2020/9524635. eCollection 2020. PMID 32832011
- [Background] Elmarakby AA, Sullivan JC. Relationship between oxidative stress and inflammatory cytokines in diabetic nephropathy. Cardiovasc Ther. 2012 Feb;30(1):49-59. doi: 10.1111/j.1755-5922.2010.00218.x. Epub 2010 Aug 16. PMID 20718759
- [Background] Sandireddy R, Yerra VG, Areti A, Komirishetty P, Kumar A. Neuroinflammation and oxidative stress in diabetic neuropathy: futuristic strategies based on these targets. Int J Endocrinol. 2014;2014:674987. doi: 10.1155/2014/674987. Epub 2014 Apr 30. PMID 24883061
- [Background] Kasznicki J, Kosmalski M, Sliwinska A, Mrowicka M, Stanczyk M, Majsterek I, Drzewoski J. Evaluation of oxidative stress markers in pathogenesis of diabetic neuropathy. Mol Biol Rep. 2012 Sep;39(9):8669-78. doi: 10.1007/s11033-012-1722-9. Epub 2012 Jun 21. PMID 22718504
- [Background] Ganesh Yerra V, Negi G, Sharma SS, Kumar A. Potential therapeutic effects of the simultaneous targeting of the Nrf2 and NF-kappaB pathways in diabetic neuropathy. Redox Biol. 2013 Aug 1;1(1):394-7. doi: 10.1016/j.redox.2013.07.005. PMID 24024177
- [Background] Sheikh, W. M. E., Alahmar, I. E., Salem, G. M., & El-Sheikh, M. A. (2019). Tumor necrosis factor alpha in peripheral neuropathy in type 2 diabetes mellitus. Egyptian Journal of Neurology, Psychiatry and Neurosurgery, 55(1), 1-7. https://doi.org/10.1186/s41983-019-0080-0
- [Background] Heidari N, Sajedi F, Mohammadi Y, Mirjalili M, Mehrpooya M. Ameliorative Effects Of N-Acetylcysteine As Adjunct Therapy On Symptoms Of Painful Diabetic Neuropathy. J Pain Res. 2019 Nov 19;12:3147-3159. doi: 10.2147/JPR.S228255. eCollection 2019. PMID 31819599
- [Background] Vallianou N, Evangelopoulos A, Koutalas P. Alpha-lipoic Acid and diabetic neuropathy. Rev Diabet Stud. 2009 Winter;6(4):230-6. doi: 10.1900/RDS.2009.6.230. Epub 2009 Dec 30. PMID 20043035
- [Background] Beeh KM, Beier J, Esperester A, Paul LD. Antiinflammatory properties of ambroxol. Eur J Med Res. 2008 Dec 3;13(12):557-62. PMID 19073395
- [Background] Su X, Wang L, Song Y, Bai C. Inhibition of inflammatory responses by ambroxol, a mucolytic agent, in a murine model of acute lung injury induced by lipopolysaccharide. Intensive Care Med. 2004 Jan;30(1):133-40. doi: 10.1007/s00134-003-2001-y. Epub 2003 Sep 20. PMID 14504727
- [Background] Xia DH, Xi L, Xv C, Mao WD, Shen WS, Shu ZQ, Yang HZ, Dai M. The protective effects of ambroxol on radiation lung injury and influence on production of transforming growth factor beta1 and tumor necrosis factor alpha. Med Oncol. 2010 Sep;27(3):697-701. doi: 10.1007/s12032-009-9271-3. Epub 2009 Jul 28. PMID 19636975
- [Background] Sunkari S, Thatikonda S, Pooladanda V, Challa VS, Godugu C. Protective effects of ambroxol in psoriasis like skin inflammation: Exploration of possible mechanisms. Int Immunopharmacol. 2019 Jun;71:301-312. doi: 10.1016/j.intimp.2019.03.035. Epub 2019 Mar 29. PMID 30933843
- [Background] Puschmann S, Engelhorn R. [Pharmacological study on the bromhexine metabolite ambroxol (author's transl)]. Arzneimittelforschung. 1978;28(5a):889-98. No abstract available. German. PMID 581987
- [Background] Schutz A, Gund HJ, Pschorn U, Aicher B, Peil H, Muller A, de Mey C, Gillissen A. Local anaesthetic properties of ambroxol hydrochloride lozenges in view of sore throat. Clinical proof of concept. Arzneimittelforschung. 2002;52(3):194-9. doi: 10.1055/s-0031-1299879. PMID 11963647
- [Background] Weiser T (2000) The secretolytic ambroxol blocks neuronal Na+channels. Soc Neurosci Abstr 454.14.
- [Background] Weiser T, Wilson N. Inhibition of tetrodotoxin (TTX)-resistant and TTX-sensitive neuronal Na(+) channels by the secretolytic ambroxol. Mol Pharmacol. 2002 Sep;62(3):433-8. doi: 10.1124/mol.62.3.433. PMID 12181417
- [Background] Weiser T. Comparison of the effects of four Na+ channel analgesics on TTX-resistant Na+ currents in rat sensory neurons and recombinant Nav1.2 channels. Neurosci Lett. 2006 Mar 13;395(3):179-84. doi: 10.1016/j.neulet.2005.10.058. Epub 2005 Nov 15. PMID 16293367
- [Background] Gaida W, Klinder K, Arndt K, Weiser T. Ambroxol, a Nav1.8-preferring Na(+) channel blocker, effectively suppresses pain symptoms in animal models of chronic, neuropathic and inflammatory pain. Neuropharmacology. 2005 Dec;49(8):1220-7. doi: 10.1016/j.neuropharm.2005.08.004. Epub 2005 Sep 21. PMID 16182323
- [Background] Pawlinski L, Krawczyk M, Fiema M, Tobor E, Kiec-Wilk B. Dual-action ambroxol in treatment of chronic pain in Gaucher Disease. Eur J Pain. 2020 May;24(5):992-996. doi: 10.1002/ejp.1538. Epub 2020 Mar 9. PMID 31994807
- [Background] Kern KU, Weiser T. Topical ambroxol for the treatment of neuropathic pain. An initial clinical observation. Schmerz. 2015 Dec;29 Suppl 3(Suppl 3):S89-96. doi: 10.1007/s00482-015-0060-y. PMID 26589711
- [Background] Mullin S, Smith L, Lee K, D'Souza G, Woodgate P, Elflein J, Hallqvist J, Toffoli M, Streeter A, Hosking J, Heywood WE, Khengar R, Campbell P, Hehir J, Cable S, Mills K, Zetterberg H, Limousin P, Libri V, Foltynie T, Schapira AHV. Ambroxol for the Treatment of Patients With Parkinson Disease With and Without Glucocerebrosidase Gene Mutations: A Nonrandomized, Noncontrolled Trial. JAMA Neurol. 2020 Apr 1;77(4):427-434. doi: 10.1001/jamaneurol.2019.4611. PMID 31930374
- [Background] Narita A, Shirai K, Itamura S, Matsuda A, Ishihara A, Matsushita K, Fukuda C, Kubota N, Takayama R, Shigematsu H, Hayashi A, Kumada T, Yuge K, Watanabe Y, Kosugi S, Nishida H, Kimura Y, Endo Y, Higaki K, Nanba E, Nishimura Y, Tamasaki A, Togawa M, Saito Y, Maegaki Y, Ohno K, Suzuki Y. Ambroxol chaperone therapy for neuronopathic Gaucher disease: A pilot study. Ann Clin Transl Neurol. 2016 Feb 2;3(3):200-15. doi: 10.1002/acn3.292. eCollection 2016 Mar. PMID 27042680